CLINICAL TRIAL: NCT04987008
Title: Risk of Ischaemic Stroke After Pulmonary Embolism in Patients With and Without Patent Foramen Ovale (29BRC21.0082)
Brief Title: Risk of Ischaemic Stroke After Pulmonary Embolism in Patients With and Without Patent Foramen Ovale
Acronym: EPIC-FOPCohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: Cohorte EPIC-FOP
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-04

CONDITIONS: Foramen Ovale, Patent
Keywords: foramen ovale, patent; stroke; pulmonary embolism
MeSH Terms: conditions — Foramen Ovale, Patent; Stroke; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
stroke's risk is increased in patients with pulmonary embolism and PFO compared to patients without PFO. Does this increased risk persist years after pulmonary embolism ?

DETAILED DESCRIPTION:
324 patients included in EPIC-FOP study (2009 to 2015) were followed annually to collect data about the recurrence of VTE, cardiovascular events and treatments.

ELIGIBILITY:
Inclusion Criteria:

* patients included in EPIC-FOP study

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 53 of the 324 EPIC-FOP patients not followed in previous PE cohort
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
stroke | pulmonary embolism (2009 to 2015) to 2021
  documented stroke

SECONDARY OUTCOMES:
TIA or stroke | pulmonary embolism (2009 to 2015) to 2021
  documented TIA or stroke
death | pulmonary embolism (2009 to 2015) to 2021
  all deaths and cardiovascular deaths
bleeding | pulmonary embolism (2009 to 2015) to 2021
  Major and clinically pertinent bleeding (ISTH classification)
VTE | pulmonary embolism (2009 to 2015) to 2021
  recurrent VTE

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - HIA, Brest
  - CHRU de Brest, Brest
  - CHIC de Quimper, Quimper

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending five years following the final study report completion.
Access Criteria: Data access request will be reviewed by the internal committee of Brest University Hospital. Requestor will be required to sign and complete a data access agreement.